CLINICAL TRIAL: NCT01862991
Title: Protocol Title: Reducing Complications and Patient Barriers in Second Trimester Abortion: Pre-Operative Effects of Mifepristone (POEM) on Dilatation and Evacuation Services
Brief Title: Pre-Operative Effects of Mifepristone on Dilation and Evacuation Services
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-05132013-108659; PF-108666 (Other Grant/Funding Number: Packard Foundation)
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Legally Induced Abortion Without Mention of Complication
Keywords: Induced Abortion; Mifepristone; Dilation and Evacuation; Cervical Preparation; Osmotic Dilators
MeSH Terms: conditions — Dilatation, Pathologic | interventions — Misoprostol; Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dilapan-Placebo (Placebo Comparator): The clinician will place 4 or 5 osmotic cervical dilators (Dilapan-S)(4mm x 65mm). The patient will be administered a placebo pill orally with juice or water by the clinician or study investigator. Patients that are over 22 weeks gestation will receive 1mg of intra-amniotic digoxin the day prior to the procedure.
  Interventions: Other: Hygroscopic cervical dilators; Drug: Misoprostol; Drug: Intra-amniotic digoxin
- Dilapan-Mifepristone (Active Comparator): The clinician will place 4 or 5 osmotic cervical dilators (Dilapan-S) (4mm x 65mm). The patient will be administered mifepristone (200mg) orally with juice or water by the clinician or study investigator.Patients that are over 22 weeks gestation will receive 1mg of intra-amniotic digoxin the day prior to the procedure.
  Interventions: Other: Hygroscopic cervical dilators; Drug: Misoprostol; Drug: Intra-amniotic digoxin; Drug: Mifepristone
- Mifepristone (Experimental): The patient will be administered mifepristone (200mg) orally with juice or water by the clinician or study investigator. Patients that are over 22 weeks gestation will receive 1mg of intra-amniotic digoxin the day prior to the procedure.
  Interventions: Drug: Misoprostol; Drug: Intra-amniotic digoxin; Drug: Mifepristone

INTERVENTIONS:
Other: Hygroscopic cervical dilators — Dilapan-S osmotic cervical dilators inserted through the internal os.
  Other Names: Dilapan-S
  Arms: Dilapan-Mifepristone; Dilapan-Placebo
Drug: Misoprostol — 400 mcg buccal misoprostol 90 pre-op
Drug: Intra-amniotic digoxin — 1mg digoxin administered intra-amniotically ~24 hours pre-op in patients that are greater than 22 weeks gestation
Drug: Mifepristone — 200 mcg Mifepristone orally
  Other Names: Danco; Mifeprex
  Arms: Dilapan-Mifepristone; Mifepristone

SUMMARY:
This research study investigates the use of a drug, mifepristone, given before second trimester abortion. Mifepristone is a medication that is approved for medical abortion during the first trimester. It also has been used prior to abortion in the early seconds trimester (14-16 weeks gestation) and for medication abortion in the second trimester (also called induction abortion). This medication has effects on the uterus that may help dilate, or open, the cervix. Abortion requires opening of the cervix to safely remove the pregnancy. Cervical dilation, or opening, is essential to both ease of completion of procedure and reducing complications that can occur. These complications include laceration, or tearing, of the cervix and perforation of the uterus (a hole made unintentionally in the muscle wall of the uterus) and are not expected to be increased in the study. Dilation of the cervix is usually achieved by placing thin rods (cervical dilators) through the cervix. These rods then absorb the moisture of the vagina and slowly expand, opening the cervix. The standard method of dilation is performed at the clinic and involves the placement of cervical dilators the day before the procedure. This procedure can be uncomfortable. A prior study showed that mifepristone reduces the number of osmotic dilators that need to be placed prior to the procedure after 19 weeks gestation. We aim to investigate mifepristone as a potential adjunct to cervical dilation or used alone, without dilators, as method of cervical preparation with the hopes of reducing barriers imposed by painful procedures and time in clinic and away from work/home that the current approach involving dilators requires.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Viable, Singleton pregnancy
* Voluntarily seeking abortion between 19 and 24 wks gestation
* Able to give informed consent and comply with study protocol
* Fluent in English or Spanish

Exclusion Criteria:

* Allergy to misoprostol or mifepristone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Santa Clara Valley Medical Center, San Jose, California
  - Stanford University Medical Center, Stanford, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dilapan-Placebo | Dilapan-Mifepristone | Mifepristone
Started | 24 | 28 | 28
Completed | 21 | 27 | 27
Not Completed | 3 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dilapan-Placebo | Dilapan-Mifepristone | Mifepristone | Total
Number analyzed (Participants) | 21 | 27 | 27 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7) | 27.5 (6) | 27 (6) | 28 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 27 | 27 | 75
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 27 | 27 | 75

OUTCOME MEASURES:

1. Primary Outcome: Procedure Time
Description: Measured as time from speculum insertion to removal
Time Frame: Intraoperative Time, Collected immediately within procedure
Measure: Median (Full Range); unit: minutes
Arm/Group | Dilapan-Placebo | Dilapan-Mifepristone | Mifepristone
Number analyzed (Participants) | 21 | 27 | 27
minutes | 13 [6 to 26] | 12 [7 to 25] | 18.5 [8 to 52]

2. Secondary Outcome: Adverse Events
Description: Uterine perforation
Time Frame: Intraoperatively and 2 weeks post operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan-Placebo | Dilapan-Mifepristone | Mifepristone
Number analyzed (Participants) | 21 | 27 | 27
Participants | 0 | 1 | 2

ADVERSE EVENTS:
Arm/Group | Dilapan-Placebo | Dilapan-Mifepristone | Mifepristone
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/27 | 2/27
Other Adverse Events (participants affected / at risk) | 1/21 | 0/27 | 5/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dilapan-Placebo (N=21) | Dilapan-Mifepristone (N=27) | Mifepristone (N=27)
Uterine Perforation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dilapan-Placebo (N=21) | Dilapan-Mifepristone (N=27) | Mifepristone (N=27)
Cervical Laceration (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No